CLINICAL TRIAL: NCT05125653
Title: Indocyanine Green Fluorescent Cholangiography and Intraoperative Angiography With Laparoscopic Cholecystectomy, a Randomized Controlled Trial
Brief Title: Indocyanine Green Fluorescent Cholangiography and Intraoperative Angiography With Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohammad Ahmad Abd-erRazik, Lecturer of General Surgery, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: AinShamsSurg2
Record Dates: First submitted 2021-10-04; First posted 2021-11-18 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Cholecystitis; Chronic Calculous Cholecystitis; Acute Calculous Cholecystitis
Keywords: Laparoscopic Cholecystectomy; Indocyanine Green Fluorescent Cholangiography; Indocyanine Green Fluorescent Angiography
MeSH Terms: conditions — Cholecystitis; Cholecystitis, Acute

STUDY DESIGN:
Intervention Model Description: 2 arms, randomized, double blinded
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIR/ICG Arm (Experimental): Indocyanine Green Fluorescent Cholangiography and Intraoperative Angiography will be done during the Laparoscopic Cholecystectomy
  Interventions: Procedure: Indocyanine Green Fluorescent Laparoscopic Cholangiography
- WL Arm (Active Comparator): Conventional white light was used for Laparoscopic Cholecystectomy
  Interventions: Procedure: White Light

INTERVENTIONS:
Procedure: Indocyanine Green Fluorescent Laparoscopic Cholangiography — Indocyanine Green Fluorescent Cholangiography
  Other Names: Indocyanine Green Fluorescent LaparoscopicCholangiography
  Arms: NIR/ICG Arm
Procedure: White Light — Performing the laparoscopic cholecystectomy and identifying the biliary structures under the conventional white light
  Other Names: WL
  Arms: WL Arm

SUMMARY:
This was a double blinded, randomized, controlled trial involved patients underwent laparoscopic cholecystectomy

DETAILED DESCRIPTION:
A double blinded, randomized, controlled trial involved patients underwent laparoscopic cholecystectomy in Ain-Shams University Specialized Hospital in the period from January 2020 till July 2021. Group A (n=60) underwent laparoscopic cholecystectomy using the usual white light, Group B (n=58) underwent laparoscopic cholecystectomy with ICG florescence cholangiography and intraoperative ICG florescence arteriography.

ELIGIBILITY:
Inclusion Criteria:

* adults (from 18 to 75 years old)
* suffering from a gall bladder disease
* with valid indication for laparoscopic cholecystectomy (e.g., calculus gall bladder with cholecystitis)
* accepted to participate in the study.

Exclusion Criteria:

* Patients with history of previous biliary surgery
* Patients with abdominal malignancy
* Patients with advanced chronic liver disease
* pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Visual identification of the biliary tree | during the procedure
  To measure the % of patients in which investigators can identify visually the extra hepatic biliary system (the CD, CBD, CHD, and any possible anomalies present), during LC.
Visual identification of the cystic artery | during the procedure
  To measure the % of patients in which investigators can identify visually the cystic artery, during LC.

SECONDARY OUTCOMES:
Visual identification of injuries | during and imediatly after the procedure (24 hours)
  To detect of incidence rate of biliary or vascular injury, visually or clinically, resulted from miss identification of the structures.
Compare operative time | during the procedure
  To compare the operative time in (minutes)
Compare blood loss | during the procedure
  To compare the operative blood loss (in cc)
Compare blood loss in cc | during the procedure
  To compare the blood loss (in cc) between the two groups.
Percentage of patients of ICG adverse reactions | Within 24 hour of the procedure
  To measure % of patients suffering off reactions related to the use of ICG (by vital data assessment, monitor patients' complaints, etc..)

CONTACTS AND LOCATIONS:
Overall Officials: M Abd-erRazik, MD, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University Hospitals - AUSH, Cairo, Egypt